CLINICAL TRIAL: NCT04459637
Title: Surveillance of COVID-19 Using Smart Wearable Devices: a Prospective Study
Brief Title: COVID-19 Surveillance Based on Smart Wearable Device
Acronym: COVID-19SWD
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guangfa Wang, Professor & MD., Peking University First Hospital
Other Study IDs: 2020055-0615
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: COVID-19 Surveillance Smart wearable device
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Asymptomatic group: Definition of asymptomatic disease:refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)
- Mild group: Definition of mild disease:refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)
- general-type group: Definition of general-type disease:refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)
- severe group: Definition of severe disease:refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)
- critical group: Definition of critical disease:refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)

SUMMARY:
This is a prospective, multi-center cohort study. 200 subjects with COVID-19will be included . Wearable device's physiological parameters and clinical data will be continually collected , the investigators aim to explore whether using smart wearable devices is useful to early alerting deterioration of COVID-19.

DETAILED DESCRIPTION:
This is a prospective cohort study. 200 subjects aged 18～75y with asymptomatic, mild, general-type COVID-19 will be recruited. The physiological parameters of wearable devices, including heart rate, sleep, blood oxygen saturation, electrocardiogram and exercise records, will be continuously collected from the day of admission / isolation to 14 days after discharge or out of quarantine. The Department of Respiratory and Critical Care of Peking University First Hospital is responsible for this research. All clinical data of patients during hospitalization will be collected including demographic characteristics, onset time, visit time, hospitalization time, symptoms, physical examination, laboratory examination, imaging characteristics, disease severity, treatment and outcome. Primary outcome is the deterioration of disease, the correlation analysis between the change of wearable device physiological parameters and the deterioration of disease determined by the traditional disease evaluation system will be used to find it whether can early alert deterioration of COVID-19.

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2020-055). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years(both 18 and 75), either gender;
2. At the time of enrollment, patients with novel coronavirus infection meeting the criteria of The New Coronavirus Pneumonia Diagnosis and Treatment Program (Seventh Edition)
3. Able to engage in daily activities;
4. Willing to participate in this research and willing to follow the research program, with the ability to sign informed consent;
5. having mobile communication equipment which can install APP of wearable device.

Exclusion Criteria:

1. Wear time of wearable devices <50% during the whole study period
2. Wearable devices have faults, missing signals or errors throughout the study period, resulting in the proportion of analyzable information <50%
3. Patients with incomplete outpatient and inpatient information and missing core information such as hospitalization / discharge time, symptoms, laboratory examination, disease progress record, etc.
4. Patients with serious underlying diseases (including serious mental diseases, mental disorders, nervous system diseases, malignant tumors, chronic liver diseases, heart failure, autoimmune diseases, chronic kidney diseases), or life expectancy less than 6 months
5. Unable to take care of themselves in daily life, unable to cooperate with medical history and data collection
6. participating in other clinical trials;
7. Pregnant women, women in puerperium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with novel coronavirus infection meeting the criteria of The New Coronavirus Pneumonia Diagnosis and Treatment Program (Seventh Edition)
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Deterioration of the condition | 30 minutes
  Deterioration of the condition: refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 7)
  1. The development from asymptomatic to mild/general-type
  2. The development from mild to general-type/severe type
  3. The development from general-type to severe/critical type
  4. The development from severe to critical type

SECONDARY OUTCOMES:
Mortality | 14days and/or 28days
  Mortality within 14days and 28days after admission
The information analysis degree, the proportion of signal loss, the proportion of wrong signal, | 30 minutes
  The information analysis degree, the proportion of signal loss, the proportion of wrong signal

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang C, Sun A, Liao J, Zhang C, Yu K, Ma X, Wang G. COVID-19 surveillance based on consumer wearable devices. Digit Health. 2024 Apr 24;10:20552076241247374. doi: 10.1177/20552076241247374. eCollection 2024 Jan-Dec. PMID 38665889